CLINICAL TRIAL: NCT05301179
Title: The Mechanistic Underpinning of Protein Quality and Quantity in Aging Skeletal Muscle: A High Sensitivity Dynamic Proteome Profiling Approach
Brief Title: Protein Quantity and Quality in Older Subjects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: National Dairy Council (Other); Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 7929
Record Dates: First submitted 2021-09-27; First posted 2022-03-29 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Aging
Keywords: protein; plant-based; dairy; aging

STUDY DESIGN:
Intervention Model Description: In a partial factorial cross-over design, subjects will be assigned to one of two protein daily intakes and complete two different levels of dietary protein quality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDA Lacto-Vegetarian/Vegan (Experimental): Subjects will receive diets containing the RDA for protein from Lacto-vegetarian and Vegan sources in different periods during the protocol.
  Interventions: Other: Protein quantity and quality
- Higher than RDA Lacto-Vegetarian/Vegan (Experimental): Subjects will receive diets containing more than the RDA for protein from Lacto-vegetarian and Vegan sources in different periods during the protocol.
  Interventions: Other: Protein quantity and quality

INTERVENTIONS:
Other: Protein quantity and quality — Participants will ingest Lacto-vegetarian and vegan diets providing different daily protein quantities. The parallel design will test for protein quantity and the cross-over design will compare the effects of the quality of the protein sources in the diet.

SUMMARY:
After the age of ~50, humans start to lose muscle mass at a rate of about 1-3% per year. However, the loss of muscle mass beyond a certain point can make it increasingly difficult to perform activities of daily living such as rising from a chair, going up and downstairs, carrying groceries, etc. A reason why muscle mass is lost with age is that skeletal muscles become less sensitive to the growth-promoting effects of physical activity and protein ingestion. This loss of sensitivity can be overcome by consuming larger amounts of protein; however, many older adults have difficulties simply consuming greater amounts of protein from whole-food sources. Therefore, the research in this study aims to investigate how different amounts and types of protein, of either a 100%-plant-based or Lacto-vegetarian (plant-based plus dairy) protein sources, affect muscle growth. This information will be important when providing information to older adults about the amount and type of protein that should be consumed by older adults to help prevent the loss of muscle mass that typically occurs with advancing age.

ELIGIBILITY:
Inclusion Criteria:

1. Be a male or female, between the ages of 65 - 80 years (inclusive)
2. Be willing and able to provide informed consent
3. Be in general good health, non-smoking
4. Have a body mass index (BMI) between 20-35 kg/m2 (inclusive)

Exclusion Criteria:

1. Use of tobacco or related products.
2. Any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements.
3. Use assistive walking devices (e.g., cane or walker)
4. History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years.
5. Significant orthopedic, cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude oral protein supplement ingestion and/or assessment of safety and study objectives.
6. Any cachexia-related condition (e.g., relating to cancer, tuberculosis or human immunodeficiency virus infection and acquired immune deficiency syndrome) or any genetic muscle diseases or disorders
7. Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation, difficulty swallowing)
8. Hypersensitivity or known allergy to any of the components in the diets.
9. Excessive alcohol consumption (>21 units/week)
10. History of bleeding diathesis, platelet or coagulation disorders, or antiplatelet/anticoagulation therapy (up to 81mg of baby aspirin per day taken as a prophylactic is permitted).
11. History of statin myalgia.
12. Personal or family history of a clotting disorder or deep vein thrombosis;
13. Concomitant use of corticosteroids, testosterone replacement therapy (ingestion, injection, or transdermal), any anabolic steroid, creatine, whey protein supplements, casein, or branched-chain amino acids (BCAAs) within 45 days prior to screening.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic proteome profiling (synthesis and breakdown) | Resulting data after two weeks following a vegan and a lacto-vegetarian diet
  Proteins from skeletal muscle samples will be extracted and fractionated by sodium dodecyl sulfate - polyacrylamide gel electrophoresis (SDS-PAGE). The gel bands corresponding to 10 discrete molecular weight regions will be excised from Coomassie blue-stained gels and digested. The peptides will be extracted from the gel for liquid chromatography-mass spectrometry (LC/MS) analysis. Protein identifications will be based on the Uniprot/Swissprot database. A visual basic application will be used to predict mass isotopomer patterns over a range of precursor body 2H2O enrichments (p) for each peptide, based on the number (n) of C-H positions in the summed amino acids in each peptide that actively incorporate 2H from body water. Fractional synthesis rates (%) of proteins will be calculated by deconvoluting the mass isotopomer pattern of newly synthesized peptide species as compared to unlabeled species and, from this, calculating the fraction of newly synthesized peptides present.
Integrated muscle protein synthesis | Integrated total protein synthesis after two weeks following a vegan and a lacto-vegetarian diet
  Participants will ingest deuterated water for two weeks when following a vegan and a lacto-vegetarian diet according to a cross-over experimental design. Skeletal muscle biopsies will be collected before and after two weeks to return the integrated muscle protein synthesis representative of two weeks. Muscle protein synthesis data will be calculated based on the incorporation of deuterated alanine in muscle proteins. Muscle samples will be prepared for gas chromatography-mass spectrometry (GC-MS) analysis of the individual amino acids. Data obtained from GC-MS will be used to calculate integrated muscle protein synthesis (%.d-1).
Whole-body protein balance | After two weeks on an experimental diet, whole body protein balance will be measured during a day visit to the lab
  Participants will report to the lab to participate in a 2-period tracer infusion-metabolic study. Using stable isotope tracers, fasting and fed protein kinetics will be assessed. Fasting protein kinetics will be assessed during a 3.5h infusion. The fed protein balance will be assessed for 4h after consumption of a test meal at three different times during the visit. Blood samples will be collected at several time-points following tracer infusion to measure tracer enrichment. The calculation of whole-body protein kinetics (protein synthesis, protein breakdown, and net protein balance) will be based on the determinations of the rate of appearance (Ra) of phenylalanine (Phe) and tyrosine into plasma and the fractional Ra of endogenous tyrosine resulting from Phe hydroxylation. For that, will be applied a 2-pool model (g of protein.h-1).

SECONDARY OUTCOMES:
Cell signaling pathways regulating protein synthesis in skeletal muscle | Acute - Fed response (2h after ingestion of a test meal - this will be measured twice during the study - the response to a vegan meal and a to lacto-vegetarian meal).
  Phosphorylation of proteins in the Akt/mTORC1 pathway measured by SDS-page electrophoresis followed by Western-blotting (Arbitrary units).
Daily plasma amino acid concentration | One day in response to 3 main meals (twice during the study - 1 day ingesting vegan meals and another day ingesting lacto-vegetarian meals)
  Plasma amino acid concentrations will be analyzed via gas chromatography-mass spectrometry using the Phenomenex EZfaast amino acid analysis kit per the manufacturer's instructions (umol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, PhD, Principal Investigator — McMaster University, Department of Kinesiology
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No